CLINICAL TRIAL: NCT00464178
Title: A Phase II Study of Bevacizumab and Bortezomib in Patients With Relapsed Refractory Multiple Myeloma
Brief Title: A Phase II Study of Bevacizumab and Bortezomib in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed early due to poor accrual
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV3502s; AVF3502s (Other: Protocol no.); 20070359 (Other: WIRB no.)
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; myeloma; relapsed myeloma; refractory myeloma; relapsed, refractory myeloma; relapsed, refractory multiple myeloma; refractory multiple myeloma; relapsed multiple myeloma; B lymphoid malignancies; Myeloma, Plasma-Cell; Myeloma Proteins; hnRNP A1; myeloma helix-destabilizing protein, mouse; IgC3kappa Jir protein, human; gamma 3 myeloma protein Jir, human; M-proteins (Myeloma); M315 myeloma protein, mouse; myeloma protein M 315, mouse; McPC603 antibody; myeloma protein McPC603 antibody; multiple myeloma M-proteins; M protein, multiple myeloma; myeloma cell activator; myeloma immunoglobulins; myeloma immunoglobulin M603; myeloma immunoglobulin S15; myeloma protein A48, mouse; A48 myeloma protein, mouse; ABPC48 myeloma protein, mouse; myeloma protein A 48, mouse; myeloma protein Dob; myeloma protein M 467; myeloma protein M467; myeloma protein MOPC 141, mouse; MOPC141 myeloma protein, mouse; myeloma protein MOPC 173; myeloma protein Rou; IgA2 myeloma protein Rou; myeloma protein TEPC15; myeloma protein T15; myeloma protein TEPC 15; myeloma protein W3129; myeloma protein WIE; myeloma-associated membrane antigen KMA; myeloma antigen KMA; MYEOV protein, human; protein 460; myeloma protein MOPC 460; TRAPPC1 protein, human; multiple myeloma protein 2, human; Wis heavy-chain disease protein, human; myeloma protein Wis, human
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib and bevacizumab (Experimental): Bortezomib will be administered at 1.3 mglm2 IVP on Days 1. 4, 8, and 11. Response will be assessed subsequent to each cycle. A total of 8 cycles would beplanned. Patients would be removed subsequent to Cycle 2. if progression of disease is documented.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered at 1.3 mglm2 IVP on Days 1. 4, 8, and 11. Response will be assessed subsequent to each cycle. A total of 8 cycles would beplanned. Patients would be removed subsequent to Cycle 2. if progression of disease is documented.
  Other Names: Bortezomib will be administered

SUMMARY:
The purpose of this study is to determine whether the combination of bevacizumab and bortezomib have increased efficacy in the treatment of relapsed/ refractory multiple myeloma.

DETAILED DESCRIPTION:
Rationale: With the identification of thalidomide as an active agent in Multiple Myeloma, the role of angiogenesis in its pathogenesis has become a subject of much investigation. Micro vessel density (neovascularization) is inversely related to prognosis in Multiple Myeloma. Response to thalidomide was felt to correlate with a decline in microvessel density (Singhal et al NEJM). While the mechanism of neovascularization is yet to be fully elucidated, a number of models have shown VEGF to play a central role.

Thalidomide has been shown to synergize with a number of agents used to treat MM, including bortezomib. (Wang et al ASH 2005) This would justify the use of other therapeutics with known antiangiogenic activity in conjunction with established antimyeloma therapies.

Bortezomib, which has the precedence of known synergy with Thalidomide and has an extremely well established optimal dose, schedule, response rate, event free survival, and overall survival would make it an excellent candidate for combination therapy with other established antiangiogenic compounds.

There have been several reports of the role of VEGF in multiple myeloma. It has been shown that multiple myeloma cells secreteVEGF, which further promotes production of IL-6 in BMSCs, as well as migration and proliferation of the tumor cells. Thus VEGF is both an autocrine growth factor and trigger of IL-6-mediated paracrine multiple myeloma cell growth. Recent reports have highlighted the major role of VEGF in multiple myeloma pathogenesis, demonstrating the VEGF also increases microvessel density in the bone marrow. VEGF also inhibits dendritic cells. Taken together, these preclinical reports make strong suggestion for the promise of VEGF targeted agents in multiple myeloma (Le Gouill et al 2004).

ELIGIBILITY:
Inclusion Criteria:

* Must have been previously diagnosed with multiple myeloma based on Durie-Salmon criteria and/or the diagnostic criteria developed by the International Myeloma Working Group (IMWG).The patient must currently require therapy for relapsed (progressive disease, defined as a 25% increase in M-protein, development of new or worsening of existing lesions or soft tissue plasmacytoma, or hypercalcemia, or relapse from CR. Or patient must have disease that is refractory to most recent therapy. Defined as less than a 50% reduction in serum paraprotein or 90% reduction in urine paraprotein.
* Must have measurable disease, defined as follows: For secretory multiple myeloma, measurable levels of monoclonal protein: greater than or equal to 0.5g/dL on electrophoresis or greater than or equal to 200mg of monoclonal light chain on a 24 hour protein electrophoresis.
* Must have had at least one prior line of therapy but no more than three prior lines of therapy.
* Must understand and voluntarily sign an informed consent form.
* Must be greater than/equal to 18 years of age at time of signing consent.
* Must be able to adhere to study visit schedule and other protocol requirements.
* Must have an ECOG performance status of 0,1or 2
* Women of Child-bearing potential (WCBP) defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive method; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study medication.
* All WCBP and all sexually active male patients must agree to use adequate methods of birth control throughout the study.

Exclusion Criteria:

* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 12 weeks
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure or left ventricular ejection fraction (LVEF) < 40% (Note: baseline evaluation of LVEF should be performed for any patient who has received >450mg/m2 of any anthracycline during prior chemotherapy.
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known CNS disease
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Known hypersensitivity to any component of bevacizumab and/or bortezomib
* Previously treated with Bortezomib and/or Bevacizumab.
* Received nitrosoureas within 3 weeks or any other chemotherapy, including thalidomide or clarithromycin, or radiation therapy before enrollment.
* Received corticosteroids (greater than 10mg/day prednisone or equivalent) within three weeks prior to enrollment.
* Received immunotherapy or antibody therapy within 8 weeks prior to enrollment.
* Received plasmapheresis within 4 weeks before enrollment.
* Had major surgery within 4 weeks before enrollment. (kyphoplasty is not considered major surgery)
* History of allergic reactions attributable to compounds containing boron or mannitol.
* Grade 3 or greater peripheral neuropathy as defined by the NCI Common Toxicity Criteria (NCI CTC version 3.0) Grade 3: Sensory loss or paresthesia interfering with ADLs. Grade 4: Permanent sensory loss that interferes with function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Siegel, MD, PhD, Principal Investigator — The Cancer Center at Hackensack University Medical Center
Locations (1):
- The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 subjects completed study during study period 6/14/2007 to 9/14/2008 at medical hospital location
Pre-assignment Details: Seven subjects were consented, six were treated and one screen failed. Of the six treated, 4 completed, one subject was taken off study because of non compliance to protocol, one withdrew
Period: Overall Study
Arm/Group | Bortezomib and Bevacizumab
Started | 6
Completed | 4
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 7 subjects were consented 6 proceeded with treatment, 4 completed study: one failed screening and one was dropped due to non-compliance with protocol, one withdrew consent
Groups:
- Drug Combination: Overall Survival (OS) - Overall Survival is Calculated at the Time of the Screening Evaluation to Death From Any Cause.
Arm/Group | Drug Combination
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Cycles to Tumor Progression (TTP)
Description: Study Schema: Bortezomib will be administered on Days 1. 4, 8, and 11. Response will be assessed subsequent to each 21-day cycle. Progression is defined using the Bladé criteria, defined progression as an increase of >25% in paraprotein or urinary light chain excretion (or marrow plasma cell percentage in the marrow
Time Frame: 18 months
Measure: Median (Full Range); unit: Cycles Prior to Tumor Progression
Arm/Group | Bortezomib and Bevacizumab
Number analyzed (Participants) | 6
Cycles Prior to Tumor Progression | 1.5 [1 to 10]

2. Primary Outcome: Overall Survival (OS) - Number of Participants Alive at Study Completion
Description: The secondary objective of this study is to assess the safely and tolerability of the combination treatment of bevacizumnab and bortezomnib. Adjustments in the dosing schedule of bortezomib would be made for patients with adequate response as per Blade criteria and continue until disease progression or 18 months
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Bortezomilb and Bevacizumab: Bortezomilb will be administered at 1.3 mglm2 IVP on Days 1. 4, 8, and 11. Response will be assessed subsequent to each cycle. A total of 8 cycles would beplanned. Patients would be removed subsequent to Cycle 2. if progression of disease is documented.
Arm/Group | Bortezomilb and Bevacizumab
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: period of study
Arm/Group | Drug Combination
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The study was terminated prior to enrollment completion and formal analysis of the primary objectives was never conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes